CLINICAL TRIAL: NCT05745779
Title: Serum Vitamin D, HbA1c and Vitamin B12 Levels in Patients With Gingivitis and Periodontitis Stages
Brief Title: Vitamin D, HbA1c and Vitamin B12 Levels in Patients
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Selcen Ozcan Bulut, Assistant professor, Nigde Omer Halisdemir University
Other Study IDs: 2022/81
Record Dates: First submitted 2023-02-03; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Serum HbA1c and Vitamin D, Vitamin B12 Values in Periodontal Diseases
Keywords: Diabetes Mellitus; Periodontitis; Risk Factors; Vitamin
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Gingivitis: 0% interdental bone loss
  Interventions: Diagnostic Test: HbA1c, Vitamin D, Vitamin B12
- Stage 1 periodontitis: 0-15% interdental bone loss
  Interventions: Diagnostic Test: HbA1c, Vitamin D, Vitamin B12
- Stage 2 Periodontitis: 15-33% interdental bone loss
  Interventions: Diagnostic Test: HbA1c, Vitamin D, Vitamin B12
- Stage 3 Periodontitis: >33% interdental bone loss with potential for additional tooth loss
  Interventions: Diagnostic Test: HbA1c, Vitamin D, Vitamin B12
- Stage 4 Periodontitis: >%33 interdental bone loss with potantial for loss of dentition
  Interventions: Diagnostic Test: HbA1c, Vitamin D, Vitamin B12

INTERVENTIONS:
Diagnostic Test: HbA1c, Vitamin D, Vitamin B12 — Serum HbA1c, Vitamin D, Vitamin B12 values of the patients who applied for gingival treatment in the last 3 months from the date of application were found from the hospital archive and serum was not taken from the patients again for the study.

SUMMARY:
Abstract Aim: to compare the serum vitamin D, HbA1c and vitamin B12 levels in patients with gingivitis and four different periodontitis stages diagnosed according to the 2017 Periodontal Disease Classification.

Materials and methods: A total of 606 (378 Female, 228 Male) patients were included in the study. The periodontal status of the patients was diagnosed with gingivitis, stage 1,2,3 and 4 periodontitis groups were formed. HbA1c, vitamin D and vitamin B12 values of the patients were compared and analyzed.

Result:

Conclusion:

DETAILED DESCRIPTION:
bstract Aim: to compare the serum vitamin D, HbA1c and vitamin B12 levels in patients with gingivitis and four different periodontitis stages diagnosed according to the 2017 Periodontal Disease Classification as determined by the American Academy of Periodontology and the European Federation of Periodontology (AAP-EFP) Materials and methods: A total of 606 (378 Female, 228 Male) patients were included in the study. The periodontal status of the patients was diagnosed with gingivitis, stage 1,2,3 and 4 periodontitis groups were formed. HbA1c, vitamin D and vitamin B12 values of the patients were compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gingivitis or periodontitis with complete periodontal diagnostic data (Gingival Index(Löe, 1967), Plaque Index(Löe, 1967), Periodontal pocket depths(PD), Clinical Attachment loss (CAL), Radiological data- Interdental Bone loss (IBL) data
* Non-smoker
* Vit D, HbA1c and B12 vit in blood on the date of application to the clinic and/or in the last 3 months. Patients with data on values were included in the study.

Exclusion Criteria:

* Patients with missing data and not allowing data use
* Smoker
* The data of pregnant and lactating patients were not included in the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-80, who applied to the clinic due to periodontal disease, and had serum HbA1c, vitamin D, vitamin B12 values in the hospital archive within 3 months from the date of clinical application.
Sampling Method: Probability Sample
Enrollment: 606 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | t0:baseline
  serum Hemoglobin A1c value
Vitamin D | t0 : baseline
  serum Vitamin D value
Vitamin B12 | t0:baseline
  serum Vitamin B12 value

CONTACTS AND LOCATIONS:
Locations (1):
- Nigde Omer Halisdemir University, Dentistry Faculty, Periodontology Department, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Derived] Bulut SO, Noyun D, Dirikan Ipci S, Cakar G. Serum vitamin D, hemoglobin A1c and vitamin B12 levels in patients with gingivitis and periodontitis stages. Biomark Med. 2024;18(9):449-457. doi: 10.1080/17520363.2024.2342236. Epub 2024 May 17. PMID 39007836